CLINICAL TRIAL: NCT05226702
Title: A Phase 1 Clinical Trial to Study the Safety and Immunogenicity of a COVAC-2 Booster Dose in Generally Healthy Adults.
Brief Title: Clinical Trial to Study the COVAC-2 Booster Dose (for COVID-19) in Generally Healthy Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Government of Canada (Other Government); Government of Saskatchewan (Other Government); Vaccine Formulation Institute (VFI) (Unknown); Seppic (Industry)
Responsible Party: Principal Investigator, Volker Gerdts, Director & CEO, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: COVAC-004
Record Dates: First submitted 2022-02-03; First posted 2022-02-07 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Double Vaccinated for COVID-19 (For Phase 1 of the Study); Acute Respiratory Syndrome Coronavirus 2 (For Phase 2 Exploratory Group)
MeSH Terms: interventions — COVAC-1 COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- COVAC-2 10 µg group (Experimental): 20 healthy adults ≥18 years of age receive the vaccine on Day 0.
  Interventions: Biological: COVAC-2
- COVAC-2 25 µg group (Experimental): 20 healthy adults ≥18 years of age receive the vaccine on Day 0
  Interventions: Biological: COVAC-2
- Placebo Control (Placebo Comparator): 20 healthy adults ≥18 years of age receive a dose of normal saline (placebo) on Day 0.
  Interventions: Biological: Saline Placebo

INTERVENTIONS:
Biological: COVAC-2 — Intramuscular vaccine against SARS-CoV-2
  Arms: COVAC-2 10 µg group; COVAC-2 25 µg group
Biological: Saline Placebo — Intramuscular injection of saline placebo
  Arms: Placebo Control

SUMMARY:
VIDO has developed a vaccine called COVAC-2.

The COVAC-2 study vaccine contains a portion of the SARS-CoV-2 spike protein, called S1. The spike protein is the part of the virus that is responsible for attaching to the surface of host cells. COVAC-2 contains a SWE adjuvant. An adjuvant is a compound that is added to a vaccine to help the vaccine produce a better immune response. The SWE adjuvant is similar to another adjuvant, MF59, that is found in influenza vaccines and MF59 containing vaccines have been given to millions of people around the world. The vaccine is expected to stimulate the body to make antibodies against the S1 protein. The antibodies will recognize the viral spike protein if the body is exposed to the virus and prevent severe COVID-19 illness. In animal studies, the immune response generated by the COVAC-2 vaccine was able to protect the vaccinated animals against a severe SARS-CoV-2 infection.

This is a Phase 1/2, placebo-controlled, observer-blind, age-stratified randomized, multicenter study to access the safety and immunogenicity of two dosing levels (10 and 25 µg S1 protein tested in parallel) administered once in healthy adults ≥18 of age who have received 2 doses of an authorized COVID-19 vaccine at least 6 months earlier. The study will also include an open-label exploratory study arm to evaluate safety and immunogenicity of a single COVAC-2 dose in previously SARS-CoV-2-infected individuals (Phase 2 only).

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy male and female adults aged 18 years or older at the time of signing the informed consent form.
* Good general health as determined by screening evaluation no greater than 30 days before injection of study vaccine.

Note: Participants who are overtly healthy as determined by medical evaluation or are considered medically stable according to the judgment of the Investigator. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 3 months prior to enrolment, and/or hospitalization within the entire study period is not anticipated. Also, the participant appears likely to be able to remain in follow-up through the end of protocol-specified period. Mild to moderate well-controlled comorbidities are allowed.

* Have received minimum of 2 doses of an authorized COVID-19 vaccine at least 4 months prior to Day 0.
* Male participant and females of child-bearing potential and heterosexually active, practice of adequate contraception for 30 days prior to injection, negative pregnancy test on the day of injection, and agreement to continue adequate contraception until 180 days after the injection.
* Written informed consent, after review of the consent form and having adequate opportunity to discuss the study with an Investigator or a qualified designee.

Exclusion Criteria:

* Presence of any febrile illness or any known or suspected acute illness on the day of immunization.
* Any condition, which in the opinion of the Investigator may make the participant inappropriate for the study.
* Clinically significant bleeding disorder (e.g., clotting factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following intramuscular injections or venipuncture.
* Receiving systemic immunomodulatory therapy or history of receiving chemotherapy in the last 5 years other than topical agents.
* Receipt of systemic glucocorticoids (a dose ≥20 mg/day prednisone or equivalent for 14 days) within 1 month, or any other cytotoxic or immunosuppressive drug within 6 months prior to injection of study vaccine.
* Cancer diagnosis in the last 5 years, excluding basal cell and squamous cell carcinoma of the skin, which are allowed.
* Presence of autoimmune disease.
* Receipt of any investigational drug within 6 months.
* Receipt of any non-COVID-19 authorized vaccines, for example influenza, within 2 weeks of receiving study dose injection.
* Receipt of any other experimental SARS-CoV-2/COVID-19 or other experimental coronavirus vaccine(s) at any time prior to or during the study. Exception: Receipt of SARS CoV 2/COVID-19 vaccines at least 4 months prior to Day 0 that were experimental at the time of their administration but are currently authorized will not lead to exclusion.
* Receipt of blood products or immunoglobulin (IVIg or IMIg) within 3 months of study entry/baseline serologic evaluation.
* Current anti-tuberculosis therapy.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study vaccine.
* Hematologic or biochemical laboratory abnormalities (blood or urine), as defined by lab normal ranges. To exclude transient abnormalities, the Investigator may repeat a test once, and if the repeat test is normal according to local reference ranges, participant may be enrolled. Abnormalities of laboratory values will not be exclusionary if considered not clinically significant by the Investigator.
* Previous (within 4 months prior to Day 0) SARS-CoV-2 infection, based on a documented positive polymerase chain reaction (PCR) test or rapid antigen test, or reported by participant or prior medical history.
* Member of the study personnel, or immediate family member or household member of the study personnel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Assessment of the safety and tolerability of COVAC-2 booster vaccine in generally healthy volunteers | Up to 365 days
  Incidence of solicited adverse events (AE) up to 7 days post-injection; unsolicited AEs up to 28 days post-injection; any clinically significant laboratory finding up to 28 days post-injection; and any serious AEs (SAEs), potential immune medicated disease (pIMDs) or COVID-19 illness up to 365 days.

SECONDARY OUTCOMES:
To assess the spike binding and neutralizing response induced by COVAC-2 booster vaccine | Up to 365 days
  Antibody response induced by COVAC-2 booster pre-injection and post injection as measured by spike protein-specific Enzyme Linked Immunosorbent Assay (ELISA), virus microneutralization and/or pseudovirus neutralization assay.
To assess the immune response induced by COVAC-2 booster vaccine, as measured by cell immune response markers up to Day 365. | Up to 365 days
  Measurement of COVAC-2 immune response by measuring cell-mediated response markers in Peripheral Blood Mononuclear Cells (PBMCs) pre- and post-injection.

OTHER OUTCOMES:
Explore the effect of the age group, number of previous COVID-19 vaccine doses and type of previous COVID-19 vaccine on immune response | Up to 365 days
  Antibody response induced by COVAC-2 booster pre-injection and post injection as measured by spike protein-specific ELISA, virus neutralization assay against variant of concern, by measuring cell-mediated response markers in Peripheral Blood Mononuclear Cells (PBMCs).

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Manna Research (Burlington North), Burlington, Ontario
  - Manna Research, Toronto, Ontario
  - Canadian Center for Vaccinology, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garg R, Liu Q, Van Kessel J, Asavajaru A, Uhlemann EM, Joessel M, Hamonic G, Khatooni Z, Kroeker A, Lew J, Scruten E, Pennington P, Deck W, Prysliak T, Nickol M, Apel F, Courant T, Kelvin AA, Van Kessel A, Collin N, Gerdts V, Koster W, Falzarano D, Racine T, Banerjee A. Efficacy of a stable broadly protective subunit vaccine platform against SARS-CoV-2 variants of concern. Vaccine. 2024 Aug 13;42(20):125980. doi: 10.1016/j.vaccine.2024.05.028. Epub 2024 May 19. PMID 38769033